CLINICAL TRIAL: NCT07095348
Title: Relationship Between Serum Xanthine Oxidase Levels and Seborrheic Keratosis
Acronym: SK-XO
Status: Completed | Type: Observational
Sponsor: Sri Nauli Dewi Lubis (Other)
Responsible Party: Sponsor-Investigator, Sri Nauli Dewi Lubis, Universitas Sumatera Utara, Universitas Sumatera Utara
Organization: Universitas Sumatera Utara (Other)
Other Study IDs: SK-XO-2024-USU
Record Dates: First submitted 2025-07-16; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Seborrheic Keratosis (SK); Oxidative Stress; Skin Aging
Keywords: Xanthine Oxidase; Reactive Oxygen Species; Skin Lesions; Benign Skin Tumor; Dermatology; Facial Hyperpigmentation; ELISA; Cross-Sectional Study; UV Exposure; Guanine Deaminase
MeSH Terms: conditions — Keratosis, Seborrheic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples were collected from venous blood of all participants to measure xanthine oxidase (XO) levels. Blood was drawn, allowed to clot, and then centrifuged to obtain the serum. The serum samples were analyzed using a Human Xanthine Oxidase ELISA Kit. No DNA was extracted, and no genetic testing was performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Seborrheic Keratosis Group: This group includes 40 participants diagnosed with seborrheic keratosis through clinical and dermoscopic examination. Venous blood was collected to measure serum xanthine oxidase (XO) levels using ELISA. Participants were between 18 and 50 years old and had no underlying systemic diseases. This group represents the case population in this observational case-control study.
  Interventions: Other: Serum Xanthine Oxidase Level Assessment
- Control Group: This group includes 40 healthy participants without seborrheic keratosis or other hyperpigmented skin lesions. They were age- and sex-matched to the case group. Blood samples were collected to determine serum XO levels using the same ELISA protocol. These individuals served as the control group for comparison of XO levels.
  Interventions: Other: Serum Xanthine Oxidase Level Assessment

INTERVENTIONS:
Other: Serum Xanthine Oxidase Level Assessment — Blood samples were collected from each participant and serum was separated by centrifugation. Serum xanthine oxidase (XO) levels were measured using a Human XO ELISA Kit (Cat No. E3495Hu) according to the manufacturer's instructions. This intervention involved no therapeutic intent and was performed for observational biomarker analysis only.

SUMMARY:
This observational study aims to examine the relationship between serum xanthine oxidase (XO) levels and seborrheic keratosis (SK), a common benign skin tumor, especially in middle-aged and older adults. The pathogenesis of SK remains unclear, but oxidative stress is believed to play a role. XO is an enzyme that contributes to the production of reactive oxygen species (ROS), which can cause oxidative damage in the skin.

A total of 80 participants will be included in the study, consisting of 40 patients diagnosed with SK and 40 healthy individuals as controls. Each participant will undergo clinical and dermoscopic examination, followed by blood sampling to measure serum XO levels using ELISA. The study will be conducted at the Dermatology and Venereology Clinic of Prof. dr. Chairuddin Panusunan Lubis Universitas Sumatera Utara Hospital from October 2023 to June 2024.

This study has been reviewed and approved by the Ethics Committee of the Faculty of Medicine, Universitas Sumatera Utara.

DETAILED DESCRIPTION:
Seborrheic keratosis (SK) is one of the most common benign skin tumors observed in dermatology practice. Although SK is not malignant, its appearance can be concerning to patients, particularly when lesions are numerous or located on visible areas such as the face. The exact cause of SK is unknown, but multiple factors such as age, genetics, ultraviolet (UV) exposure, and oxidative stress have been implicated.

This observational study is designed to investigate the potential association between serum xanthine oxidase (XO) levels and the presence of SK. XO is a pro-oxidant enzyme involved in purine metabolism that generates reactive oxygen species (ROS), including superoxide and hydrogen peroxide. These ROS may play a role in oxidative stress, which is thought to contribute to various skin aging processes and possibly to benign epidermal proliferative conditions like SK.

A total of 80 participants are included in the study: 40 patients diagnosed with SK and 40 healthy controls without SK. Participants are between 18 and 50 years old and recruited from the dermatology outpatient clinic. All subjects undergo clinical and dermoscopic examination for confirmation of diagnosis. Blood samples are collected from all participants, and serum XO levels are measured using a validated enzyme-linked immunosorbent assay (ELISA) technique.

Strict inclusion and exclusion criteria are applied to minimize confounding variables, such as the presence of other dermatologic conditions, systemic illnesses, or recent antioxidant treatment. This protocol is aimed at providing foundational data to explore the biochemical basis of SK and the potential involvement of oxidative mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 50 years
* Willing to participate and sign informed consent
* Able to undergo dermatologic and dermoscopic examination
* For case group: diagnosed with seborrheic keratosis
* For control group: no clinical or dermoscopic evidence of seborrheic keratosis

Exclusion Criteria:

* History or presence of other hyperpigmentation skin lesions (e.g., lentigo solaris)
* Diagnosed with systemic diseases such as diabetes mellitus, cardiovascular disease, hepatitis, HIV/AIDS, gout, or renal impairment
* Taking medications that affect oxidative stress biomarkers
* Pregnant or breastfeeding women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants aged 18 to 50 years recruited from the dermatology outpatient clinic, including patients with seborrheic keratosis and healthy individuals without skin lesions.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Serum Xanthine Oxidase Concentration Measured by ELISA in Patients With and Without Seborrheic Keratosis | Single measurement during study visit (cross-sectional)
  This outcome measures the serum concentration of xanthine oxidase (XO) using a Human Xanthine Oxidase ELISA Kit (Cat. No E3495Hu) in participants aged 18-50 years. The concentration is expressed in ng/mL. Blood samples are collected from both seborrheic keratosis (SK) patients and healthy control participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. dr. Chairuddin Panusunan Lubis Universitas Sumatera Utara Hospital, Medan, North Sumatra, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to serum xanthine oxidase (XO) levels, age, sex, and occupational category will be shared. No personally identifiable information will be included.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data and supporting documents will be available starting January 1, 2026, for a period of 5 years or upon reasonable request while the study findings remain relevant.
Access Criteria: Qualified researchers affiliated with academic or research institutions may request access to the data by contacting the corresponding author. Requests must include a brief research proposal and intended use. Access will be granted via secure data transfer following ethics committee review if necessary.